CLINICAL TRIAL: NCT02126566
Title: Phase 2 Study of Multiclear Treatment for Striae Distensae - A Pilot Study
Brief Title: Multiclear Treatment for Striae Distensae - A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/00518
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Striae Distensae
Keywords: striae distensiae
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Administration of light therapy - measurement of results before and after therapy
  Interventions: Device: Administration of light therapy - measurement of results before and after therapy

INTERVENTIONS:
Device: Administration of light therapy - measurement of results before and after therapy

SUMMARY:
Striae distensae is a common skin condition that rarely causes significant medical problems. However, it often results in a considerable amount of distress to those with the condition. Various modalities of treatments have been used for striae distensae but few have led to satisfactory results.

More recently, newer techniques such as pulsed dye laser and radiofrequency devices have been used with modest results. There is still, however, paucity of data using light therapy for the treatment of this condition. Blue light therapy using the Multiclear device has been used successfully in the treatment of acne. In contrast, there is little data to suggest its use in the management of striae distensae.

We aim to study the effects of blue light on the treatment of striae distensae and whether this can be used safely to manage this condition.

DETAILED DESCRIPTION:
Patients will receive twice weekly blue light treatment with the Multiclear device. The first treatment dose will be 75mJ/cm2 ( Minimum Effective Dose;MED) for all patients. If no erythema develops, the subsequent treatment dose can be increased by 0.5 MED. If mild to moderate erythema develops, the same dose (i.e. 1 MED) will be used.If severe erythema/ blisters develop, treatment will be stopped and the patient wil be invited one week later and treatment will be offered at 50% of the last dose.

During the first consultation, patients will be assessed for the presence of striae distensae (SD). Duration and previous treatments of SD will be recorded. The width of the widest striae and the length of the longest straie will be measured at baseline and after 2 months of treatment. Photographs will be taken at baseline and post treatment. These will be evaluated by dermatologists who will be blinded (i.e. details of which photographs are pre or post treatment will not be given). Subjective scores will be used (Very good to excellent; >75%, Good; 51-75%, Moderate; 26-50%, Minimal to no improvement; <25%) Participants will also be given a feedback form to rate any improvements noted and any side effects experienced.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female subjects
2. Patients above 21 years
3. Patients who are able to attend follow up regularly

Exclusion Criteria:

1. Patients with other co-existing dermatoses
2. Patients with epilepsy/ who are pregnant
3. Patients with previous intolerable treatment to blue light
4. Patients treated with blue light within the last six months

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction in Striae | 2 months
  The width of the widest striae and the length of the longest straie will be measured at baseline and after 2 months of treatment. Photographs will be taken at baseline and post treatment. These will be evaluated by dermatologists who will be blinded (i.e. details of which photographs are pre or post treatment will not be given). Subjective scores will be used (Very good to excellent; >75%, Good; 51-75%, Moderate; 26-50%, Minimal to no improvement; <25%)
  Participants will also be given a feedback form to rate any improvements noted and any side effects experienced.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore